CLINICAL TRIAL: NCT01220063
Title: CLINICAL MULTICENTER STUDY OF PHASE II AND RADIOBIOLOGY ASSESSING Hypofractionated Stereotactic Radiotherapy With Irinotecan (Campto) IN THE TREATMENT OF LIVER METASTASIS AND / OR PULMONARY, Unoperated or Recurrent After Surgery of a Colorectal Cancer
Brief Title: RSHF in Colorectal Cancer
Acronym: RS CAMPTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/9-R
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: RSHF; Irinotecan; Colorectal Cancer; metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Radiation; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation + Irinotecan (Other): Irinotecan will be administered :
  - 40 mg/m² in serum physiologique during 30 to 90 min at D1 and D8 of radiotherapy
  Radiotherapy (RSHF) will be administered :
  * at D1, D3, D8 and D10
  * 48 Gy, 12 Gy by fractions twice a week
  Interventions: Radiation: Radiation; Drug: Irinotecan

INTERVENTIONS:
Radiation: Radiation — 10 Gy for 4 times (total 40 Gy)
  Other Names: RSHF
Drug: Irinotecan — 40 mg/m² : Day 1 and day 8
  Other Names: Campto

SUMMARY:
The purpose of this study is to study stereotactic radiotherapy with a dose of 40 Gy in 4 fractions over 2 weeks with concomitant 40 mg/m2 of irinotecan (1st and 3rd irradiation session).

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Social Insurance
* Performance Index <2
* Life expectancy> 6 months
* adenocarcinoma colorectal (histologically proven)
* Metastases (inoperable or recurrent after surgery),
* hepatic localization and / or lung (up to 3 if one organ metastasis or 3 in total if the two bodies are metastatic). The largest diameter of the metastasis will < ou = 6cm for the liver, < or = 6 cm for the lung. If multiple metastases, the sum of their maximum diameter is 6cm < ou = the liver, < ou = 6 cm for the lung.
* Lesion (s) measurable (s) and evaluable (s)
* CT less than 3 weeks
* Patients must have received at least one prior chemotherapy regimen containing 5FU

  • Patients may have received one or more lines of chemotherapy including irinotecan.
* bilirubin <1.5 x ULN
* AST and ALT <5x ULN
* neutrophils> 1.5x109 / L, platelets> 100x109 / L, hemoglobin> 9 g / dL
* TP, TCA Normal (only for patients treated with a permanent implant)
* Informed consent signed.

Exclusion Criteria:

* contraindication to the administration of irinotecan.
* History of radiotherapy in the thoraco-abdominal-cons indicating further irradiation.
* History of other invasive cancer treated in a period of less than 5 years (basal cell carcinoma and non-invasive cervical excepted)
* Metastatic disease diffuse or more than three metastases in the liver and / or lung during the natural history of disease (excluding any patient is having a complete radiological response on several metastases although 1-3 residual after treatment ( s) medical (at)).
* Location (s) tumor (s) = CTV to less than 12 mm laterally or less than 15 mm in the cranio-caudal, stomach, small intestine, esophagus, trachea, bronchi of right and left pulmonary arteries and right and left.
* Pregnancy or breastfeeding.

  - Lack of means or refusal to use effective contraception for men or women of childbearing age.
* Any other concomitant experimental treatment.
* Any other concurrent anticancer therapy, immunotherapy or hormonal therapy.
* Monitoring impossible because of psychological, sociological or because of geographical distance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-10-19 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
tumor response accoording to recist criteria | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: RIO EMMANUEL, MD, Study Director — INSTITUT DE CANCEROLOGIE DE L'OUEST
Locations (6):
- France (6):
  - Hôpital Saint André, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Berard, Lyon
  - Centre hospitalier Lyon Sud, Lyon
  - Hôpital la Source, Orléans
  - Centre René Gauducheau, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No